

IRB ID: Pro20150001531 Approval Date: 4/30/2015 Expiration Date:

RUTGERS
New Jersey Medical School

Department of Anesthesiology
Rutgers, The State University of New Jersey
185 South Orange Ave, MSBE538b
Newark, NJ 07103

p.973 972-5007 f.973 972-0582

# Informed Consent Form-

Study Title: The Effects of Antenatal and Perinatal Education of Labor Analgesia Options on Maternal Anxiety, Labor Analgesia, and Maternal Satisfaction with Labor Analgesia

You are being asked to participate in a research study that is being conducted by the Department of Anesthesiology/New Jersey Medical School at the Rutgers University.

# Purpose of the study:

The purpose of this study is to learn how we can better educate our pregnant patients about the options open to them for pain relief during labor. If you decide to participate you will be one of approximately 100 subjects.

### What will be done?

You will receive some educational materials regarding the options for pain relief during labor. After you deliver your baby you will be asked to complete a 23 question paper survey, which will take 15-20 minutes to complete. The survey includes questions about whether you received the educational material on a visit to the obstetrician, your pain management preference prior to labor experience, method of delivery and your satisfaction with your pain control. After you complete the questionnaire, we will record your responses on a data sheet. We expect the study to last about two years. Participation in this study is voluntary. The only alternative to this study is not to participate.

#### Risks or discomforts:

There are no known anticipated risks from taking part in this study. If you feel uncomfortable with a question, you can skip that question or withdraw from the study altogether. If you decide to quit at any time before you have finished the questionnaire, your answers will NOT be recorded.

### Benefits of this study:

There is no direct benefit to you for participating in this study. You will be contributing to knowledge about patient education and patient satisfaction.

#### Confidentiality:

Your responses will be kept strictly confidential. The paper/digital data will be stored in secure computer and a hard copy will be stored in a locked filing cabinet after it is entered. Your personal identifiers (such as name, address) will not be stored with data from your survey. We will not collect any personal identifying information about you and all answers will be confidential. The paper data or hard copy will be destroyed once all data has been entered into the data base. Only the investigators will have access to the data.

RUTGERSAPPROVED

PI: Antonio Gonzalez -Fiol, MD

Title: The Effects of Antenatal and Perinatal Education of Labor Analgesia Options on Maternal An: Maternal Satisfaction with Labor Analgesia

IRB ID: Pro20150001531 Approval Date: 4/30/2015 Expiration Date:

# Compensation:

You will not be compensated for completing the study.

### Withdrawal:

Your participation is voluntary; you are free to withdraw your participation from this study at any time. If you do not want to continue, you may turn in a blank survey. You also may choose to skip any questions that you do not wish to answer.

# How the findings will be used:

The results of the study will be used to help the investigators learn what are the educational needs of our patients and how can we improve patient satisfaction. The results from the study may be presented at an educational meeting attended by anesthesiologists, and the results might be published in a Medical Journal.

### Contact information:

If you have concerns or questions about this research study, please contact Dr. Antonio Gonzalez at 973 972-5255 or the study coordinator Catherine Schoenberg at 973 972-7477.

If you have questions about your rights as a research subject, please contact the IRB Director at (973)-972-3608 Newark.

By beginning the survey, you acknowledge that you have read this information and agree to participate in this research, with the knowledge that you are free to withdraw your participation at any time without penalty.